CLINICAL TRIAL: NCT05380999
Title: The Training and Validation Study: Development of a Red Blood Cells Based Blood Test for Early Detection of Lung Cancer
Brief Title: The Red Blood Cells Based Blood Test for Lung Cancer EARLY Detection
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Peking Union Medical College Hospital (Other); Shanghai Chest Hospital (Other); Guangzhou Panyu Central Hospital (Other); My-BioMed Technology （Guangzhou） Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: GL2022-LC001
Record Dates: First submitted 2022-04-24; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Red Blood Cells; Methylation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pulmonary nodules (diameter ≤3cm) plan to diagnosis benign and malignant: Patients with pulmonary nodules (diameter ≤3cm) plan to use biopsy or surgery or treatment to diagnosis benign and malignant.
  Interventions: Diagnostic Test: Methylation tests of nucleic acids extracted from mature red blood cells (RBCs)

INTERVENTIONS:
Diagnostic Test: Methylation tests of nucleic acids extracted from mature red blood cells (RBCs) — Up to 15 ml of peripheral blood will be collected from each subject, and the blood specimen will be processed to isolate mature red blood cells and extract the DNA and RNA from RBCs. DNA and RNA methylation will be tested by next-generation sequencing (NGS).

SUMMARY:
This study plan to enroll 852 patients with pulmonary nodules smaller than 3 cm in diameter, whose DNA and RNA will be extracted from mature red blood cells isolated from peripheral blood. The DNA 5-methylcytosine(5-mC) and RNA 2'-O-methylation information will be acquired by NGS and Nm Judge Universally sequencing (NJU-Seq), which will be used to establish models to distinguish patients with benign and malignant nodule in the training group and further evaluated in the validation group. The pathological results will be acquired after surgery or biopsy as standard in the study.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, cohort study and seeks to enroll 852 participants with pulmonary nodules smaller than 3 cm in diameter from 4 hospitals in China.

Each participant pulmonary nodule is ≤30mm as assessed by CT scanning, nodule is suspected to be malignant, and plan to use biopsy or surgery for diagnosis or treatment within 60 days.Their blood samples, CT scan data, and clinical data will be collected at each visit and tissues will be collected when participants who receive pneumonectomy or percutaneous lung biopsy.

Each subject will analysis DNA and RNA methylation in nucleic acids extracted from mature red blood cells isolated from peripheral blood by next-generation sequencing (NGS) . A proprietary algorithm will be used to identify the modification sites and pattern for differentiating the benign and malignant pulmonary nodules. Sensitivity and specificity of the different methylation panels will be to evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary nodule is ≤3cm;
2. Subjects suspected of lung cancer;
3. Diagnosis or treatment by biopsy or surgery within 60 days;
4. Signed informed consent.

Exclusion Criteria:

1. History of malignant tumors;
2. Received anti-tumor therapy;
3. Can't collect the histopathological results or the pathological results are metastatic cancer;
4. Can't obtain detection information of red blood cells;
5. Pregnancy or lactating female；
6. Other situations not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The pulmonary nodule is ≤30mm as assessed by imaging; nodules were suspected to be malignant,
  2. Plan to use biopsy or surgery for diagnosis or treatment within 60 days.
Sampling Method: Probability Sample
Enrollment: 852 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-03-29 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the RBCs-based blood test for differentiating benign and malignant pulmonary nodules diameter less than 3 cm using DNA methylation analysis by NGS. | 3 years
Specificity of the RBCs-based blood test for differentiating benign and malignant pulmonary nodules diameter less than 3 cm using DNA methylation analysis by NGS. | 3 years
Positive predictive value (PPV) of the RBCs-based blood test for differentiating benign and malignant pulmonary nodules diameter less than 3 cm using DNA methylation analysis by NGS. | 3 years
Negative predictive value (NPV) of the RBCs-based blood test for differentiating benign and malignant pulmonary nodules diameter less than 3 cm using DNA methylation analysis by NGS. | 3 years

SECONDARY OUTCOMES:
Sensitivity of the RBCs-based methylation assay in the invasion of malignant pulmonary nodules. | 3 years
Specificity of the RBCs-based methylation assay in the invasion of malignant pulmonary nodules. | 3 years
Area under curve (AUC) of receiver operating characteristic curve (ROC) in the model established in this study will compare with that of Mayo Clinic and Veterans Affairs models. | 3 years
Sensitivity in the model established in this study will compare with that of Mayo Clinic and Veterans Affairs models. | 3 years
Specificity in the model established in this study will compare with that of Mayo Clinic and Veterans Affairs models. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School

IPD SHARING:
Plan to Share IPD: Undecided